CLINICAL TRIAL: NCT02694640
Title: Peers Promoting Exercise Adoption and Maintenance Among Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: National Cancer Institute (NCI) (NIH); American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Bernardine Pinto, Associate Dean, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 042015; 5R01CA183849-05 (NIH)
Record Dates: First submitted 2016-02-12; First posted 2016-02-29 (Estimated); Results first posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Exercise; Physical activity; Community volunteers; Peer mentors; Peer coaches; Social support; Exercise maintenance
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Reach Plus (Experimental): In Months 1-3, participants in this group will receive the previously tested telephone counseling for exercise. RTR volunteers or "coaches" will be asked to contact participants by telephone weekly over 3 months (12 calls). In months 4-9, participants will no longer receive calls from RTR coaches and will be encouraged to use the heart rate monitors and pedometers during exercise. Participants will continue to complete their exercise logs and receive feedback reports from study staff.
  Interventions: Behavioral: Reach Plus
- Reach Plus Phone (Experimental): In Months 1-3, participants in this group will receive the previously tested telephone counseling for exercise. RTR volunteers or "coaches" will be asked to contact participants by telephone weekly over 3 months (12 calls). In months 4-9, these participants will have the opportunity to continue to receive support calls from their coach. Participants will also continue to complete their exercise logs and receive feedback reports from study staff.
  Interventions: Behavioral: Reach Plus Phone
- Reach Plus Message (Experimental): In Months 1-3, participants in this group will receive the previously tested telephone counseling for exercise. RTR volunteers or "coaches" will be asked to contact participants by telephone weekly over 3 months (12 calls). In months 4-9, participants will receive messages by email or text to motivate, prompt and reinforce continued exercise. Participants will also continue to complete their exercise logs and receive feedback reports from study staff.
  Interventions: Behavioral: Reach Plus Message

INTERVENTIONS:
Behavioral: Reach Plus — In Months 1-3, participants in this group will receive the previously tested telephone counseling for exercise. RTR volunteers or "coaches" will be asked to contact participants by telephone weekly over 3 months (12 calls). In months 4-9, participants will no longer receive calls from RTR coaches and will be encouraged to use the heart rate monitors and pedometers during exercise. Participants will continue to complete their exercise logs and receive feedback reports from study staff.
  Arms: Reach Plus
Behavioral: Reach Plus Phone — In Months 1-3, participants in this group will receive the previously tested telephone counseling for exercise. RTR volunteers or "coaches" will be asked to contact participants by telephone weekly over 3 months (12 calls). In months 4-9, these participants will have the opportunity to continue to receive support calls from their coach. Participants will also continue to complete their exercise logs and receive feedback reports from study staff.
  Arms: Reach Plus Phone
Behavioral: Reach Plus Message — In Months 1-3, participants in this group will receive the previously tested telephone counseling for exercise. RTR volunteers or "coaches" will be asked to contact participants by telephone weekly over 3 months (12 calls). In months 4-9, participants will receive messages by email or text to motivate, prompt and reinforce continued exercise. Participants will also continue to complete their exercise logs and receive feedback reports from study staff.
  Arms: Reach Plus Message

SUMMARY:
Exercise adoption enhances well-being and recovery from breast cancer. Researchers trained American Cancer Society volunteers to provide exercise counseling to breast cancer survivors and the survivors increased their exercise in the short-term. This RCT examines the effects of three maintenance conditions on survivors' exercise participation at longer follow-ups. The cost-effectiveness of the three groups will be examined to guide implementation of this peer mentoring approach in community-based organizations.

DETAILED DESCRIPTION:
The current study, a randomized controlled trial (RCT), represents the next step of the efforts to to extend the research on physical activity to the community setting; community volunteers will deliver the intervention, thereby making physical activity interventions much more accessible to survivors. In partnership with the National American Cancer Society office (Atlanta, GA) and Reach To Recovery (RTR) programs in North Carolina, South Carolina, and Georgia, researchers at the University of South Carolina's College of Nursing will share skills, experience and resources to examine the effects of RTR coaches offering a theoretically-based 3-month exercise program among 150 breast cancer survivors to increase moderate-to-vigorous physical activity (MVPA) followed by self-monitoring (i.e. exercise logs) and feedback reports in Months 4-9 (Reach Plus), monthly phone calls from RTR coaches, self monitoring and feedback reports in Months 4-9 (Reach Plus Message) or weekly email/text messages, self-monitoring and feedback reports in Months 4-9 (Reach Plus Message). In this three group study, researchers will assess survivors' exercise, fatigue, mood, quality of life, and self-reported physical functioning at baseline, 3, 9 and 12 months. The costs of the methods vary and data on costs will be collected to guide the selection of maintenance strategies for dissemination. If the results are promising, researchers will proceed with a dissemination trial wherein the large network of RTR volunteers can expand the scope of their services to benefit breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

Women aged 21 years or over will be eligible if they:

* Have been diagnosed in the past 5 years with Stage 0-3 breast cancer.
* Are able to read and speak English.
* Are ambulatory.
* Are sedentary (i.e., do not meet recommendations for moderate-intensity PA [30 minutes/ day or more for at least 5 days/ week] or vigorous-intensity PA [20 minutes/day or more for at least 3 days/week]
* Are able to walk unassisted.
* Have access to a telephone.

Exclusion Criteria:

Women with:

* More advanced disease (Stage 4).
* Medical or psychiatric problems (e.g., substance abuse, coronary artery disease, peripheral vascular disease, diabetes, and orthopedic problems) that may interfere with protocol adherence will not be included.
* Participants will be asked to provide consent for medical chart review to extract disease and treatment variables. Eligible participants will obtain medical clearance from their physicians.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernardine M Pinto, PhD, Principal Investigator — University of South Carolina - College of Nursing
Locations (1):
- University of South Carolina, College of Nursing, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pinto BM, Dunsiger SI, Kindred MM, Mitchell S. Physical Activity Adoption and Maintenance Among Breast Cancer Survivors: A Randomized Trial of Peer Mentoring. Ann Behav Med. 2022 Aug 2;56(8):842-855. doi: 10.1093/abm/kaab078. PMID 34436552
- [Derived] Pinto BM, Dunsiger SI, Kindred MM, Mitchell S. Mediators of physical activity maintenance during a 12-month randomized controlled trial among breast Cancer survivors. J Behav Med. 2023 Oct;46(5):745-756. doi: 10.1007/s10865-023-00402-0. Epub 2023 Mar 9. PMID 36892780
- [Derived] Pinto BM, Dunsiger SI, Kindred MM, Mitchell S. Peer mentoring for physical activity adoption and maintenance among breast cancer survivors: moderators of physical activity outcomes. J Cancer Surviv. 2023 Aug;17(4):1211-1220. doi: 10.1007/s11764-021-01162-z. Epub 2022 Jan 7. PMID 34994945

RESULTS

PARTICIPANT FLOW:
Groups:
- Reach Plus: In Months 1-3, participants in this group will receive the previously tested telephone counseling for exercise. Reach to Recovery volunteers (RTR) or "coaches" will be asked to contact participants by telephone weekly over 3 months (12 calls). In months 4-9, participants will no longer receive calls from RTR coaches and will be encouraged to use the heart rate monitors and pedometers during exercise. Participants will continue to complete their exercise logs and receive feedback reports from study staff.
  Reach Plus: In Months 1-3, participants in this group will receive the previously tested telephone counseling for exercise. RTR volunteers or "coaches" will be asked to contact participants by telephone weekly over 3 months (12 calls). In months 4-9, participants will no longer receive calls from RTR coaches and will be encouraged to use the heart rate monitors and pedometers during exercise. Participants will continue to complete their exercise logs and receive feedback reports from study staff.
- Reach Plus Phone: In Months 1-3, participants in this group will receive the previously tested telephone counseling for exercise. Reach to Recovery (RTR) volunteers or "coaches" will be asked to contact participants by telephone weekly over 3 months (12 calls). In months 4-9, these participants will have the opportunity to continue to receive support calls from their coach. Participants will also continue to complete their exercise logs and receive feedback reports from study staff.
  Reach Plus Phone: In Months 1-3, participants in this group will receive the previously tested telephone counseling for exercise. RTR volunteers or "coaches" will be asked to contact participants by telephone weekly over 3 months (12 calls). In months 4-9, these participants will have the opportunity to continue to receive support calls from their coach. Participants will also continue to complete their exercise logs and receive feedback reports from study staff.
- Reach Plus Message: In Months 1-3, participants in this group will receive the previously tested telephone counseling for exercise. Reach to Recovery (RTR) volunteers or "coaches" will be asked to contact participants by telephone weekly over 3 months (12 calls). In months 4-9, participants will receive messages by email or text to motivate, prompt and reinforce continued exercise. Participants will also continue to complete their exercise logs and receive feedback reports from study staff.
  Reach Plus Message: In Months 1-3, participants in this group will receive the previously tested telephone counseling for exercise. RTR volunteers or "coaches" will be asked to contact participants by telephone weekly over 3 months (12 calls). In months 4-9, participants will receive messages by email or text to motivate, prompt and reinforce continued exercise. Participants will also continue to complete their exercise logs and receive feedback reports from study staff.
Period: Overall Study
Arm/Group | Reach Plus | Reach Plus Phone | Reach Plus Message
Started | 55 | 53 | 53
Completed | 48 | 43 | 35
Not Completed | 7 | 10 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reach Plus | Reach Plus Phone | Reach Plus Message | Total
Number analyzed (Participants) | 55 | 53 | 53 | 161
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 44 | 35 | 37 | 116
  >=65 years | 11 | 18 | 16 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.09 (9.12) | 58.62 (11.01) | 56.17 (12.31) | 57.33 (10.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 53 | 53 | 161
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 1 | 4
  Not Hispanic or Latino | 52 | 53 | 52 | 157
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 15 | 3 | 9 | 27
  White | 40 | 49 | 42 | 131
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 55 | 53 | 53 | 161

OUTCOME MEASURES:

1. Primary Outcome: Physical Activity
Description: Through interviewer - administered Seven Day Activity Recall
Time Frame: 9 and 12 months
Population: All analyses were run on the intent to treat sample with all randomized participants included in the analysis
Measure: Mean (Standard Deviation); unit: min/week
Arm/Group | Reach Plus | Reach Plus Phone | Reach Plus Message
Number analyzed (Participants) | 55 | 53 | 53
min/week
  9 Months | 145.83 (153.89) | 159.86 (155.19) | 172.94 (110.83)
  12 Months | 120.81 (111.58) | 137.16 (139.31) | 135.00 (105.27)
Statistical Analysis 1: Comparison: Reach Plus vs Reach Plus Phone vs Reach Plus Message; A series of longitudinal mixed effects models with subject-specific intercepts were used to examine between-group differences in mean min/week of self reported moderate-to-vigorous physical activity (MVPA); Test type: Superiority — The study was powered to detect significant between-group differences in mean min/week MVPA at follow-up; p < .05, Regression, Linear — No adjustment for multiple comparisons was made; effect size = .11 — Effect size refers to between-group difference at follow-up

2. Primary Outcome: Min/Week Objectively Measured Moderate-to-vigorous Physical Activity
Description: Minutes per week of at least moderate intensity activity as measured by accelerometer (GT3X)
Time Frame: 9 and 12 months
Population: All analysis was conducted on the intent to treat sample with all randomized participants included in the analysis
Measure: Mean (Standard Deviation); unit: min/week
Arm/Group | Reach Plus | Reach Plus Phone | Reach Plus Message
Number analyzed (Participants) | 55 | 53 | 53
min/week
  9 months | 46.43 (73.28) | 82.17 (161.47) | 54.62 (88.13)
  12 months | 61.90 (82.11) | 68.75 (177.43) | 49.95 (67.62)
Statistical Analysis 1: Comparison: Reach Plus vs Reach Plus Phone vs Reach Plus Message; Test type: Superiority; p < .05, Regression, Linear; effect size = .09

3. Secondary Outcome: Breast Cancer Quality of Life
Description: Assessed via the Functional Assessment of Cancer Therapy Scale - Breast (FACT-B) Sub-scales scored: Physical well-being, social/family well-being, emotional well-being, functional well-being and other breast cancer related statements. Scale ranges from 0-148 with higher scores indicating higher quality of life.
Time Frame: Change at 9 and 12 months
Population: Analysis was conducted on the intent to treat sample with all randomized participants included in the analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reach Plus | Reach Plus Phone | Reach Plus Message
Number analyzed (Participants) | 55 | 53 | 53
score on a scale
  9 months | 24.72 (3.47) | 24.86 (3.63) | 24.76 (2.93)
  12 months | 24.66 (3.19) | 24.88 (3.36) | 25.12 (2.29)

4. Secondary Outcome: Fatigue
Description: Assessed via the Functional Assessment of Cancer Therapy Scale - Fatigue (FACT-F). This scale ranges from 0-52. Higher values indicate better functioning (or lower fatigue).
Time Frame: Score at 9 and 12 months
Population: Analysis was conducted on the intent to treat sample with all randomized participants included in the analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reach Plus | Reach Plus Phone | Reach Plus Message
Number analyzed (Participants) | 55 | 53 | 53
score on a scale
  9 months | 40.91 (8.64) | 42.02 (9.52) | 41.79 (7.31)
  12 months | 41.33 (8.78) | 41.66 (7.79) | 41.35 (7.60)

5. Secondary Outcome: Mood
Description: Assessed via the Profile of Mood States (POMS). Higher scores indicated a greater mood disturbance. Scale ranges from 0-28.
Time Frame: Score at 9 and 12 months
Population: Analysis was conducted on the intent to treat sample with all randomized participants included in the analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reach Plus | Reach Plus Phone | Reach Plus Message
Number analyzed (Participants) | 55 | 53 | 53
score on a scale
  9 months | 8.52 (23.38) | 8.82 (33.89) | 7.71 (17.20)
  12 months | 7.73 (23.91) | 5.12 (20.93) | 7.59 (18.48)

ADVERSE EVENTS:
Time Frame: Each participant was in the trial for 12 months.
Arm/Group | Reach Plus | Reach Plus Phone | Reach Plus Message
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/53 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/53 | 0/53
Other Adverse Events (participants affected / at risk) | 2/55 | 0/53 | 2/53
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reach Plus (N=55) | Reach Plus Phone (N=53) | Reach Plus Message (N=53)
Fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Participant fell while walking.
Pulled muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Patient pulled a muscle and required ice and ibuprofen to reduce the pain.
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) — Patient reported being out of breath during her walk.

LIMITATIONS AND CAVEATS:
Limitations include limited generalizability of the findings. Further, retention rates differed by treatment condition.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/40/NCT02694640/Prot_SAP_000.pdf